CLINICAL TRIAL: NCT02031367
Title: Efficacy of Platelet Rich Plasma vs. Corticosteroid Injections for Treating Greater
Brief Title: Efficacy of Platelet Rich Plasma vs. Corticosteroid Injections for Treating Greater Trochanteric Pain Syndrome
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: C.R.Darnall Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, MAJ Aaron Williams, Family/Sports Medicine Staff, Family Medicine Residency Center, C.R.Darnall Army Medical Center
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: GTPS PRP VS Steroid
Record Dates: First submitted 2014-01-08; First posted 2014-01-09 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Greater Trochanteric Pain Syndrome
MeSH Terms: interventions — Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Corticosteroid (Active Comparator)
  Interventions: Drug: Triamcinolone Acetonide
- Platelet Rich Plasma (Experimental)
  Interventions: Other: Platelet Rich Plasma

INTERVENTIONS:
Drug: Triamcinolone Acetonide — Corticosteroid arm
  Arms: Corticosteroid
Other: Platelet Rich Plasma — Platelet Rich Plasma
  Other Names: PRP
  Arms: Platelet Rich Plasma

SUMMARY:
The object of this study is to compare the effect of PRP versus Corticosteroid injection on pain in patients with Greater Trochanteric Pain Syndrome up to 12 months after treatment. It is believed that PRP will be as good as corticosteroids for short term pain relief, and will produce longer lasting pain reduction.

DETAILED DESCRIPTION:
The purpose of this study is to compare the efficacy of Platelet Rich Plasma (PRP) injections versus Corticosteroid injections in treating patients that have failed noninvasive management for Greater Trochanteric Pain Syndrome (GTPS). We will be comparing in both the short term (0-6 months) and in the long term (6-12 months). It will be a Double-Blinded Randomized Clinical Trial. Patients with GTPS will be randomly assigned to either the Corticosteroid group or PRP group. There will be a total of 50 participants enrolled with 25 in each group. The PRP group will receive 3 mL of autologous plasma injection into the area of tendinopathy utilizing ultrasound guidance. One (1) injection per month will be administered for a total of three (3) injections. The Corticosteroid Group will receive 2.0 mL's injection of lidocaine and 40mg of Triamcinolone into the area of tendinopathy utilizing ultrasound guidance on their first injection. They will then receive 2.0 mL's of 1% lidocaine and 3.0 mL's of 0.9% Sodium Chloride per month for a total of three (3) injections. Both groups will be referred to physical therapy. Participant's pain will be assessed using a Visual Analog Scale (VAS) and the Nonarthritic Hip Score (NHS) for function at the beginning of the treatment and then again at 1, 3, 6, 9, and 12 months after the initial injection.

ELIGIBILITY:
Inclusion Criteria:

* Males or females ages 18 and older.
* Active duty soldiers and military health care beneficiaries.
* Have lateral hip pain in the region of the greater trochanter for at least 6 weeks and have done physical therapy.
* Reproducible pain on palpation of the greater trochanteric region.
* Tendinopathy diagnosed with ultrasound. The criteria is as follows: a well-defined hypoechoic area with partial tear or complete tendon rupture that is suggestive of a tendon tear. A hyperechoic intratendinous area with posterior acoustic shadowing suggestive of a calcification, or both

Exclusion Criteria:

* Received corticosteroid for the condition in last 6 months.
* History of surgery in affected hip.
* Allergy to Lidocaine.
* Allergy to Corticosteroid.
* Unavailable for follow up by telephone for 12 months after initial injection.
* Patients with broken skin or skin infections immediately overlying the area to be injected.
* Patients with complete tears of the gluteal tendons with retraction of the muscle and or tendon, as determined by ultrasound.
* If they are pregnant or planning on becoming pregnant during the study time. Because of the physiologic changes during pregnancy we cannot predict how Corticosteroids will affect the mother and the infant. Also, this will increase stress to an already immunocompromised state.
* Have not attended formal physical therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-03; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Pain | 1 year
  Will use Visual Analog scale to measure overalll pain at 0, 1, 3, 6, 9, and 12 months of both groups to compare efficacy of both treatments.

SECONDARY OUTCOMES:
Functional outcomes | 1 year
  Will use Nonarthritic Hip score at 0, 1, 3, 6, 9, and 12 months to evaluate overall function of the patients between the two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Carl R. Darnall Army Medical Center, Fort Hood, Texas, United States

REFERENCES:
- [Background] Williams BS, Cohen SP. Greater trochanteric pain syndrome: a review of anatomy, diagnosis and treatment. Anesth Analg. 2009 May;108(5):1662-70. doi: 10.1213/ane.0b013e31819d6562. PMID 19372352
- [Background] Bird PA, Oakley SP, Shnier R, Kirkham BW. Prospective evaluation of magnetic resonance imaging and physical examination findings in patients with greater trochanteric pain syndrome. Arthritis Rheum. 2001 Sep;44(9):2138-45. doi: 10.1002/1529-0131(200109)44:93.0.CO;2-M. PMID 11592379
- [Background] Strauss EJ, Nho SJ, Kelly BT. Greater trochanteric pain syndrome. Sports Med Arthrosc Rev. 2010 Jun;18(2):113-9. doi: 10.1097/JSA.0b013e3181e0b2ff. PMID 20473130
- [Background] Brinks A, van Rijn RM, Willemsen SP, Bohnen AM, Verhaar JA, Koes BW, Bierma-Zeinstra SM. Corticosteroid injections for greater trochanteric pain syndrome: a randomized controlled trial in primary care. Ann Fam Med. 2011 May-Jun;9(3):226-34. doi: 10.1370/afm.1232. PMID 21555750
- [Background] El-Husseiny M, Patel S, Rayan F, Haddad F. Gluteus medius tears: an under-diagnosed pathology. Br J Hosp Med (Lond). 2011 Jan;72(1):12-6. doi: 10.12968/hmed.2011.72.1.12. PMID 21240111
- [Background] Lachiewicz PF. Abductor tendon tears of the hip: evaluation and management. J Am Acad Orthop Surg. 2011 Jul;19(7):385-91. doi: 10.5435/00124635-201107000-00001. PMID 21724917
- [Background] Del Buono A, Papalia R, Khanduja V, Denaro V, Maffulli N. Management of the greater trochanteric pain syndrome: a systematic review. Br Med Bull. 2012 Jun;102:115-31. doi: 10.1093/bmb/ldr038. Epub 2011 Sep 4. PMID 21893483
- [Background] Lustenberger DP, Ng VY, Best TM, Ellis TJ. Efficacy of treatment of trochanteric bursitis: a systematic review. Clin J Sport Med. 2011 Sep;21(5):447-53. doi: 10.1097/JSM.0b013e318221299c. PMID 21814140
- [Background] Labrosse JM, Cardinal E, Leduc BE, Duranceau J, Remillard J, Bureau NJ, Belblidia A, Brassard P. Effectiveness of ultrasound-guided corticosteroid injection for the treatment of gluteus medius tendinopathy. AJR Am J Roentgenol. 2010 Jan;194(1):202-6. doi: 10.2214/AJR.08.1215. PMID 20028924
- [Background] Mautner K, Colberg RE, Malanga G, Borg-Stein JP, Harmon KG, Dharamsi AS, Chu S, Homer P. Outcomes after ultrasound-guided platelet-rich plasma injections for chronic tendinopathy: a multicenter, retrospective review. PM R. 2013 Mar;5(3):169-75. doi: 10.1016/j.pmrj.2012.12.010. Epub 2013 Feb 9. PMID 23399297
- [Background] van Ark M, Zwerver J, van den Akker-Scheek I. Injection treatments for patellar tendinopathy. Br J Sports Med. 2011 Oct;45(13):1068-76. doi: 10.1136/bjsm.2010.078824. Epub 2011 May 3. PMID 21543346
- [Background] Connell DA, Bass C, Sykes CA, Young D, Edwards E. Sonographic evaluation of gluteus medius and minimus tendinopathy. Eur Radiol. 2003 Jun;13(6):1339-47. doi: 10.1007/s00330-002-1740-4. Epub 2002 Nov 23. PMID 12764651
- [Background] Fearon AM, Scarvell JM, Cook JL, Smith PN. Does ultrasound correlate with surgical or histologic findings in greater trochanteric pain syndrome? A pilot study. Clin Orthop Relat Res. 2010 Jul;468(7):1838-44. doi: 10.1007/s11999-009-1174-2. Epub 2009 Nov 26. PMID 19941093
- [Background] Bijur PE, Silver W, Gallagher EJ. Reliability of the visual analog scale for measurement of acute pain. Acad Emerg Med. 2001 Dec;8(12):1153-7. doi: 10.1111/j.1553-2712.2001.tb01132.x. PMID 11733293
- [Background] Christensen CP, Althausen PL, Mittleman MA, Lee JA, McCarthy JC. The nonarthritic hip score: reliable and validated. Clin Orthop Relat Res. 2003 Jan;(406):75-83. doi: 10.1097/01.blo.0000043047.84315.4b. PMID 12579003